CLINICAL TRIAL: NCT00337662
Title: Predicting Response to Risperidone Treatment Through Identification of Early-onset of Antipsychotic Drug Action in Schizophrenia.
Brief Title: Efficacy Study of Early Onset of Antipsychotic Drug Action in Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10769; F1D-US-HGMN (Other: Eli Lilly and Company); NCT00373321 (obsolete NCT alias)
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2010-02

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Olanzapine; Risperidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- 1 (Experimental): Olanzapine for Not Early Onset response (NEO) patients
  Interventions: Drug: olanzapine
- 2 (Active Comparator): Risperidone for Not Early Onset response (NEO) patients
  Interventions: Drug: risperidone
- 3 (Active Comparator): Risperidone for Early Onset response (EO) patients
  Interventions: Drug: risperidone

INTERVENTIONS:
Drug: olanzapine — 10-20 milligrams (mg), oral, daily, 10 weeks.
  Other Names: LY170053; Zyprexa
  Arms: 1
Drug: risperidone — 2-6 mg, oral, daily, for 10 weeks.
  Arms: 2
Drug: risperidone — 2-6 mg, oral, daily, 10 weeks
  Arms: 3

SUMMARY:
The current study has been designed to address the significance of early onset of response prospectively in patients treated with an atypical antipsychotic.

ELIGIBILITY:
Inclusion Criteria:

* Patients must demonstrate acute psychopathologic severity criteria and be at least moderately ill.
* Patients must have experienced an exacerbation of their illness within the previous 2 weeks.
* Patients in whom a switch to another antipsychotic medication is acutely indicated.

Exclusion Criteria:

* Patients who are deemed nonresponsive to risperidone or olanzapine.
* Patients who have been hospitalized for greater than 2 weeks immediately prior to Visit 1.
* Patients having received olanzapine or risperidone in the past 30 days.
* Treatment with clozapine within 1 year prior to Visit 1.
* Diagnosis of substance-induced psychosis by Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) criteria within 7 days of Visit 1 (or at any time during the study), or confirmed on clinical grounds within 72 hours subsequent to Visit 1 (or at any time during the study).
* A diagnosis of Parkinson's disease, dementia-related psychosis, or related disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 628 (Actual)
Dates: Start 2006-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (34):
- United States (31):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Little Rock, Arkansas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Escondido, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Garden Grove, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Glendale, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., National City, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Orange, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Diego, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Ana, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Washington D.C., District of Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fort Lauderdale, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hialeah, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chicago, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Paducah, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lake Charles, Louisiana
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Boston, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jackson, Mississippi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kansas City, Missouri
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Omaha, Nebraska
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Clementon, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cedarhurst, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Olean, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Staten Island, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toledo, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rapid City, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Memphis, Tennessee
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portsmouth, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond, Virginia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kirkland, Washington
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires, Argentina
- Russia (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Khot'kovo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow

REFERENCES:
- [Derived] Chen L, Phillips G, Johnston J, Kinon BJ, Ascher-Svanum H, Kollack-Walker S, Succop P, Naber D. The relationship, structure and profiles of schizophrenia measurements: a post-hoc analysis of the baseline measures from a randomized clinical trial. BMC Psychiatry. 2011 Dec 28;11:203. doi: 10.1186/1471-244X-11-203. PMID 22204569
- [Derived] Fijal BA, Stauffer VL, Kinon BJ, Conley RR, Hoffmann VP, Witte MM, Zhao F, Houston JP. Analysis of gene variants previously associated with iloperidone response in patients with schizophrenia who are treated with risperidone. J Clin Psychiatry. 2012 Mar;73(3):367-71. doi: 10.4088/JCP.10m06507. Epub 2011 Jul 12. PMID 21813073
- [Derived] Ascher-Svanum H, Nyhuis AW, Stauffer V, Kinon BJ, Faries DE, Phillips GA, Schuh K, Awad AG, Keefe R, Naber D. Reasons for discontinuation and continuation of antipsychotics in the treatment of schizophrenia from patient and clinician perspectives. Curr Med Res Opin. 2010 Oct;26(10):2403-10. doi: 10.1185/03007995.2010.515900. PMID 20812791
- [Derived] Kinon BJ, Chen L, Ascher-Svanum H, Stauffer VL, Kollack-Walker S, Zhou W, Kapur S, Kane JM. Early response to antipsychotic drug therapy as a clinical marker of subsequent response in the treatment of schizophrenia. Neuropsychopharmacology. 2010 Jan;35(2):581-90. doi: 10.1038/npp.2009.164. PMID 19890258
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study Period I was the screening period prior to enrollment. Study Period II was a 2-week open-label lead-in period of risperidone 2-6mg/day, at which time determination of early onset status was determined. Study Period III was a 10-week, double-blind therapy period.
Groups:
- NEO-OLZ: Olanzapine for not early onset response (NEO) patients. Olanzapine: 10-20 mg, oral, daily for 10 weeks
- NEO-RIS: Risperidone for not early onset response (NEO) patients. Risperidone: 2-6 mg, oral, daily for 10 weeks
- EO-RIS: Risperidone for early onset response (EO) patients. Risperidone: 2-6 mg, oral, daily for 10 weeks
- Risperiodone Open-Label Lead-In: All patients completed a 2-week open-label risperidone lead-in period. This group contains all patients who started Study Period II.
  Risperidone: 2-6 mg, oral, daily
Period: Study Period II
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS | Risperiodone Open-Label Lead-In
Started | 0 | 0 | 0 | 628
Completed | 0 | 0 | 0 | 522
Not Completed | 0 | 0 | 0 | 106
Not completed — Lost to Follow-up | 0 | 0 | 0 | 35
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 20
Not completed — Adverse Event | 0 | 0 | 0 | 16
Not completed — Physician Decision | 0 | 0 | 0 | 13
Not completed — Entry Criteria Not Met | 0 | 0 | 0 | 6
Not completed — Protocol Violation | 0 | 0 | 0 | 6
Not completed — Lack of Efficacy | 0 | 0 | 0 | 7
Not completed — Sponsor Decision | 0 | 0 | 0 | 2
Not completed — Parent/Caregiver Decision | 0 | 0 | 0 | 1
Period: Study Period III
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS | Risperiodone Open-Label Lead-In
Started | 186 | 192 | 144 | 0
Completed | 126 | 134 | 100 | 0
Not Completed | 60 | 58 | 44 | 0
Not completed — Lost to Follow-up | 14 | 16 | 14 | 0
Not completed — Withdrawal by Subject | 18 | 14 | 12 | 0
Not completed — Adverse Event | 9 | 10 | 8 | 0
Not completed — Protocol Violation | 3 | 8 | 2 | 0
Not completed — Physician Decision | 6 | 5 | 0 | 0
Not completed — Entry Criteria Not Met | 4 | 1 | 3 | 0
Not completed — Lack of Efficacy | 4 | 4 | 2 | 0
Not completed — Parent/Caregiver Decision | 0 | 0 | 2 | 0
Not completed — Sponsor Decision | 1 | 0 | 1 | 0
Not completed — Clinical Relapse | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS | Total
Number analyzed (Participants) | 186 | 192 | 144 | 522
Age Continuous [Mean (Standard Deviation); unit: years] | 41.84 (10.92) | 41.87 (11.34) | 41.83 (10.88) | 41.85 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 76 | 58 | 200
  Male | 120 | 116 | 86 | 322
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 2 | 1 | 4
  Asian | 3 | 0 | 0 | 3
  Black or African American | 88 | 92 | 54 | 234
  White | 80 | 80 | 74 | 234
  Hispanic | 14 | 18 | 15 | 47
Region of Enrollment [Number; unit: participants]
  United States | 173 | 176 | 130 | 479
  Argentina | 4 | 5 | 9 | 18
  Russian Federation | 9 | 11 | 5 | 25
Diagnosis [Number; unit: participants]
  Schizophrenia/Schizophreniform Disorder | 140 | 144 | 114 | 398
  Schizoaffective Bipolar Disorder | 31 | 25 | 21 | 77
  Schizoaffective Depression | 15 | 23 | 9 | 47
Abnormal Involuntary Movement Scale - Non-Global Total Score [Mean (Standard Deviation); unit: units on a scale] — A 12-item instrument assesses observed abnormal movements in different parts of body. Ten items are scored in a 5-point scale (0 = none/normal, 4 = severe) which evaluates abnormal movements in three main anatomic areas (orofacial area, extremities, and trunk). Two items are yes/no questions regarding dentures. Total scores range from 0 to 42.
  units on a scale | 0.67 (1.82) | 0.49 (1.48) | 0.44 (1.38) | 0.54 (1.58)
Barnes Akathisia Rating Scale Total Score [Mean (Standard Deviation); unit: units on a scale] — Evaluates akathisia associated with use of antipsychotic medications, includes objective and subjective component plus global impression rating for overall disorder. Components rated on scale of 0 to 3 for objective and subjective items and 0 to 5 for global clinical assessment, for total score of 0 (absence of akathisia) to 11 (severe akathisia).
  units on a scale | 0.80 (1.81) | 0.95 (1.97) | 0.54 (1.64) | 0.78 (1.83)
Modified Simpson-Angus Scale [Mean (Standard Deviation); unit: units on a scale] — Measures neuroleptic-induced parkinsonism. Total score consists of the sum of 10 items: 7 items (items 1, 3, 4, 7, 8, 9, 10) rated on a 4-point severity scale where 0=normal and 4=extreme, and 3 items (items 2, 5, 6) rated on a 2-point severity scale where 0=normal and 2=definitely abnormal/present. The total score ranges from 0 to 34.
  units on a scale | 0.12 (0.29) | 0.14 (0.29) | 0.13 (0.82) | 0.13 (0.50)
Montgomery-Asberg Depression Rating Scale (MADRS) - Total Score [Mean (Standard Deviation); unit: units on a scale] — Measures the overall severity of depressive symptoms. The MADRS has a 10-item checklist. Items are rated on a scale of 0-6, for a total score range of 0 (low severity of depressive symptoms) to 60 (high severity of depressive symptoms).
  units on a scale | 13.52 (7.98) | 12.49 (8.44) | 7.29 (6.07) | 11.42 (8.09)
Positive and Negative Syndrome Scale (PANSS) - Negative Subscale [Mean (Standard Deviation); unit: units on a scale] — Assesses negative symptoms associated with schizophrenia. 7 items make up the Negative scale (ex. blunted affect, emotional withdrawal, poor rapport, and passive/apathetic social withdrawal). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total Negative Subscale scores range from 7 to 49.
  units on a scale | 21.18 (4.96) | 20.94 (5.30) | 15.83 (3.90) | 19.62 (5.36)
Positive and Negative Syndrome Scale (PANSS) - Positive Subscale [Mean (Standard Deviation); unit: units on a scale] — Assesses positive symptoms associated with schizophrenia. 7 items make up the Positive scale (ex. delusions, conceptual disorganization, and hallucinatory behavior). Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Total Positive Subscale scores range from 7 to 49.
  units on a scale | 21.50 (4.49) | 20.95 (4.65) | 15.37 (3.97) | 19.61 (5.13)
Positive and Negative Syndrome Scale (PANSS) - Total Score [Mean (Standard Deviation); unit: units on a scale] — Assesses the positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. The scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). The sum of the 30 items is defined as the PANSS total score and ranges from 30 to 210.
  units on a scale | 84.91 (13.81) | 84.05 (14.81) | 61.67 (12.85) | 78.21 (17.24)

OUTCOME MEASURES:

1. Primary Outcome: Changes From Study Period II Baseline (Week 0) to Weeks 3, 4, 6, 8, and 12 in Positive and Negative Syndrome Scale (PANSS) Total Score in Early Onset Response and Not Early Onset Response-Risperidone Patients
Description: Assesses positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. Scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Sum of 30 items is PANSS total score and ranges from 30 to 210. Change = time point - single-blind baseline (Week 0).
Time Frame: Weeks 0, 3, 4, 6, 8, 12
Population: Intention to treat for patients with both baseline and any postbaseline assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NEO-RIS | EO-RIS
Number analyzed (Participants) | 189 | 138
units on a scale
  Change from Week 0 to Week 3 | -11.90 (1.15) | -30.80 (1.23)
  Change from Week 0 to Week 4 | -14.81 (1.16) | -32.53 (1.24)
  Change from Week 0 to Week 6 | -16.23 (1.26) | -32.90 (1.36)
  Change from Week 0 to Week 8 | -18.10 (1.31) | -34.10 (1.43)
  Change from Week 0 to Week 12 | -18.62 (1.38) | -35.09 (1.50)
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p < 0.001, Mixed Effects Model Repeated Measures — Between-group p-values for each baseline to post-baseline visit were the same, p<0.001

2. Secondary Outcome: Changes From Study Period III Baseline (Week 2) to Weeks 3, 4, 6, 8, and 12 in Positive and Negative Syndrome Scale Total Score in Not Early Onset Response-Risperidone and Not Early Onset Response-Olanzapine Patients
Description: Assesses positive symptoms, negative symptoms, and general psychopathology specifically associated with schizophrenia. Scale consists of 30 items. Each item is rated on a scale from 1 (symptom not present) to 7 (symptoms extremely severe). Sum of 30 items is PANSS total score and ranges from 30 to 210. Change = time point - double-blind baseline (Week 2).
Time Frame: Weeks 2, 3, 4, 6, 8, 12
Population: Intention to treat patients with both baseline and postbaseline assessment
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | NEO-RIS | NEO-OLZ
Number analyzed (Participants) | 189 | 179
units on a scale
  Change from Week 2 to Week 3 | -6.94 (0.82) | -5.85 (0.84)
  Change from Week 2 to Week 4 | -9.82 (0.86) | -9.67 (0.88)
  Change from Week 2 to Week 6 | -11.25 (0.98) | -13.06 (1.02)
  Change from Week 2 to Week 8 | -13.13 (1.00) | -14.73 (1.04)
  Change from Week 2 to Week 12 | -13.53 (1.13) | -17.02 (1.16)
Statistical Analysis 1: Comparison: NEO-RIS vs NEO-OLZ; Test type: Superiority or Other; p = 0.266, Mixed-Effects Model Repeated-Measures — Change from Week 2 to Week 3 p-value
Statistical Analysis 2: Comparison: NEO-RIS vs NEO-OLZ; Test type: Superiority or Other; p = 0.884, Mixed-Effects Model Repeated-Measures — Change from Week 2 to Week 4 p-value
Statistical Analysis 3: Comparison: NEO-RIS vs NEO-OLZ; Test type: Superiority or Other; p = 0.151, Mixed-Effects Model Repeated-Measures — Change from Week 2 to Week 6 p-value
Statistical Analysis 4: Comparison: NEO-RIS vs NEO-OLZ; Test type: Superiority or Other; p = 0.216, Mixed-Effects Model Repeated-Measures — Change from Week 2 to Week 8 p-value
Statistical Analysis 5: Comparison: NEO-RIS vs NEO-OLZ; Test type: Superiority or Other; p = 0.020, Mixed-Effects Model Repeated-Measures — Change from Week 2 to Week 12 p-value

3. Secondary Outcome: The Number of Participants in the Early Onset (EO) and Not Early Onset-Risperidone (NEO-RIS) Groups Who Show a 20% or Greater Reduction in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The number of participants who experienced a 20% or greater reduction in their PANSS Total score during the 12 weeks they were on risperidone.
Time Frame: Week 0 to Week 12
Population: Total number of patients having nonmissing values at both baseline (last of visit 1 - visit 2) and post baseline (last of visit 5 - visit 9) visits.
Measure: Number; unit: participants
Arm/Group | NEO-RIS | EO-RIS
Number analyzed (Participants) | 189 | 138
participants
  >=20% Reduction - Yes | 94 | 119
  >=20% Reduction - No | 95 | 19
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p < 0.001, Fisher Exact

4. Secondary Outcome: The Number of Participants in the Not Early Onset-Risperidone (NEO-RIS) and Not Early Onset-Olanzapine (NEO-OLZ) Groups Who Show a 20% or Greater Reduction in Positive and Negative Syndrome Scale (PANSS) Total Score
Description: The number of not early onset participants who experienced a 20% or greater reduction in PANSS Total Score at any time during the 12 weeks of combined Study Period II and Study Period III.
Time Frame: Week 0 to Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | NEO-RIS | NEO-OLZ
Number analyzed (Participants) | 189 | 179
participants
  >=20% Reduction - Yes | 94 | 94
  >=20% Reduction - No | 95 | 85
Statistical Analysis 1: Comparison: NEO-RIS vs NEO-OLZ; Test type: Superiority or Other; p = 0.604, Fisher Exact

5. Secondary Outcome: Number of Participants in the Early Onset and Not Early Onset-Risperidone Groups Who Show a 50% or Greater Reduction in Positive and Negative Syndrome Scale (PANSS) Total Score From Baseline or Meet 'a Priori' Specified Criteria for Remission
Description: 'a priori' specified criteria for remission defined as a score of 3 (mild), 2 (minimal), or 1 (absent) on all of the following 8 PANSS items: delusions, conceptual disorganization, hallucinatory behavior, unusual thought content, mannerisms and posturing, blunted effect, passive/apathetic withdrawal, lack of spontaneity and flow of conversation.
Time Frame: Week 0 to Week 12
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | NEO-RIS | EO-RIS
Number analyzed (Participants) | 189 | 138
participants
  >=50% Reduction - Yes | 67 | 87
  >=50% Reduction - No | 122 | 51
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p < 0.001, Fisher Exact

6. Secondary Outcome: Number of Participants in the Not Early Onset-Risperidone and Not Early Onset-Olanzapine Groups Who Show a 50% or Greater Reduction in Positive and Negative Syndrome Scale Total Score From Baseline or Meet 'a Priori' Specified Criteria for Remission
Description: as for outcome 5
Time Frame: Week 2 to Week 12
Population: Total number of patients having nonmissing values at both baseline (last of visit 3 - visit 4) and post baseline (last of visit 5 - visit 9) visits.
Measure: Number; unit: participants
Arm/Group | NEO-RIS | NEO-OLZ
Number analyzed (Participants) | 189 | 179
participants
  >=50% Reduction - Yes | 67 | 67
  >=50% Reduction - No | 122 | 112
Statistical Analysis 1: Comparison: NEO-RIS vs NEO-OLZ; Test type: Superiority or Other; p = 0.745, Fisher Exact

7. Secondary Outcome: Number of Participants With Psychiatric Hospitalizations in the Early Onset and Not Early Onset-Risperidone Groups
Description: Psychiatric Hospitalizations were measured by the Modified Schizophrenia Care and Assessment Program Health Questionnaire (SCAP-HQ) from which it could be determined the number of patients with a psychiatric episode that required an overnight stay in a hospital.
Time Frame: Week 2 to Week 12
Population: as for outcome 6
Measure: Number; unit: participants
Arm/Group | NEO-RIS | EO-RIS
Number analyzed (Participants) | 184 | 137
participants
  Required overnight stay in hospital: Yes | 9 | 10
  Required overnight stay in hospital: No | 175 | 127
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p = 0.474, Fisher Exact

8. Secondary Outcome: Vital Signs - Mean Change From Baseline to 10 Week Endpoint in Body Mass Index
Description: Body mass index is an estimate of body fat based on body weight divided by height squared. Change = Endpoint minus baseline.
Time Frame: Week 2 to Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kilogram per square meter
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Number analyzed (Participants) | 179 | 188 | 139
kilogram per square meter
  Baseline | 29.97 (8.03) | 31.05 (8.04) | 31.13 (8.77)
  Change from Baseline | 0.63 (1.38) | 0.43 (1.45) | 0.10 (1.19)
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p = 0.034, ANOVA — P-values (Change from Baseline) are based on Type III sums of squares from ANOVA model: change = group pooled investigator
Statistical Analysis 2: Comparison: NEO-OLZ vs NEO-RIS; Test type: Superiority or Other; p = 0.125, ANOVA — [p-value comment as in outcome 8, analysis 1]

9. Secondary Outcome: Number of Participants With Treatment-Emergent Abnormal Fasting Laboratory Analytes Reported in >=2% of All Participants
Description: Number of participants who experienced abnormal fasting laboratory values at any time during Study Period III. Laboratory reference ranges are dependent on the patient's gender, origin, and age.
Time Frame: Week 2 to Week 12
Population: Total number of patients with the lab test at baseline and post-baseline.
Measure: Number; unit: participants
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Number analyzed (Participants) | 179 | 188 | 139
participants
  Low total bilirubin | 5 | 3 | 2
  High creatine phosphokinase | 6 | 1 | 5
  High creatinine | 2 | 4 | 3
  High hemoglobin A1c | 6 | 7 | 2
  Low sodium | 4 | 4 | 4
  High prolactin | 7 | 8 | 7
Statistical Analysis 1: Comparison: NEO-OLZ vs NEO-RIS vs EO-RIS; Test type: Superiority or Other; p > 0.05, Fisher Exact — All comparisons between EO-RIS and NEO-RIS and between NEO-RIS and NEO-OLZ had p-values greater than 0.05

10. Secondary Outcome: Mean Change From Baseline to 10 Week Endpoint in Extrapyramidal Symptoms as Measured by the Modified Simpson-Angus Scale
Description: Measures neuroleptic-induced parkinsonism. Total score consists of the sum of 10 items: 7 items (items 1, 3, 4, 7, 8, 9, 10) rated on a 4-point severity scale where 0=normal and 4=extreme, and 3 items (items 2, 5, 6) rated on a 2-point severity scale where 0=normal and 2=definitely abnormal/present. The total score ranges from 0 to 34.
Time Frame: Week 2 to Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Number analyzed (Participants) | 168 | 173 | 133
units on a scale | -0.06 (0.27) | -0.03 (0.26) | -0.02 (0.16)
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p = 0.355, ANOVA; p-value is from ANOVA with treatment and pooled investigator in the model
Statistical Analysis 2: Comparison: NEO-OLZ vs NEO-RIS; Test type: Superiority or Other; p = 0.244, ANOVA; p-value is from ANOVA with treatment and pooled investigator in the model

11. Secondary Outcome: Mean Change From Baseline to 10 Week Endpoint in Extrapyramidal Symptoms as Measured by the Barnes Akathisia Rating Scale - Total Score
Description: Evaluates akathisia associated with use of antipsychotic medications, includes objective and subjective component plus global impression rating for overall disorder. Components rated on scale of 0 to 3 for objective and subjective items and 0 to 5 for global clinical assessment, for total score of 0 (absence of akathisia) to 11 (severe akathisia).
Time Frame: Week 2 to Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Number analyzed (Participants) | 168 | 174 | 133
units on a scale | -0.31 (1.99) | -0.13 (2.04) | -0.24 (1.38)
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p = 0.998, ANOVA; P-value is from ANOVA with treatment and pooled investigator in the model
Statistical Analysis 2: Comparison: NEO-OLZ vs NEO-RIS; Test type: Superiority or Other; p = 0.505, ANOVA; P-value is from ANOVA with treatment and pooled investigator in the model

12. Secondary Outcome: Mean Change From Baseline to 10 Week Endpoint in Extrapyramidal Symptoms as Measured by the Abnormal Involuntary Movement Scale (AIMS)- Non-Global Total Score
Description: A 12-item instrument assesses observed abnormal movements in different parts of body. Ten items are scored in a 5-point scale (0 = none/normal, 4 = severe) which evaluates abnormal movements in three main anatomic areas (orofacial area, extremities, and trunk). Two items are yes/no questions regarding dentures. Total scores range from 0 to 42.
Time Frame: Week 2 to Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Number analyzed (Participants) | 168 | 173 | 132
units on a scale | -0.38 (1.73) | 0.11 (2.07) | -0.16 (1.27)
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p = 0.266, ANOVA; P-value is from ANOVA with treatment and pooled investigator in the model
Statistical Analysis 2: Comparison: NEO-OLZ vs NEO-RIS; Test type: Superiority or Other; p = 0.015, ANOVA; P-value is from ANOVA with treatment and pooled investigator in the model

13. Secondary Outcome: Vital Signs - Mean Change From Baseline to 10 Week Endpoint in Sitting Pulse Rate
Description: Changes from Study Period III baseline to endpoint in sitting pulse rate. Change = Endpoint minus baseline.
Time Frame: Week 2 and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Number analyzed (Participants) | 179 | 188 | 139
beats per minute
  Baseline | 80.49 (11.57) | 80.84 (12.06) | 77.90 (11.02)
  Change from Baseline | -0.98 (11.81) | -2.52 (11.50) | -0.94 (12.82)
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p = 0.140, ANOVA — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: NEO-OLZ vs NEO-RIS; Test type: Superiority or Other; p = 0.181, ANOVA — [p-value comment as in outcome 8, analysis 1]

14. Secondary Outcome: Vital Signs - Change From Baseline to 10 Week Endpoint in Standing Diastolic Blood Pressure
Description: Change from Study Period III baseline to endpoint in standing blood pressure. Change = Endpoint minus baseline.
Time Frame: Week 2 and Week 12
Population: Total number of patients having nonmissing values at both baseline (last of visit 3 - visit 4) and post baseline (last of visit 5- visit 9) visits.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Number analyzed (Participants) | 176 | 184 | 137
mm Hg
  Baseline | 78.69 (10.01) | 78.57 (10.68) | 80.29 (10.65)
  Change from Baseline | 1.01 (10.79) | -0.20 (9.96) | -1.73 (8.92)
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p = 0.254, ANOVA — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: NEO-OLZ vs NEO-RIS; Test type: Superiority or Other; p = 0.299, ANOVA; P-values (Change from Baseline) are based on Type III sums of squares from ANOVA model: change = group pooled investigator

15. Secondary Outcome: Vital Signs - Change From Baseline to 10 Week Endpoint in Standing Mean Arterial Pressure
Description: Change from Study Period III baseline to endpoint in standing mean arterial pressure. Change = Endpoint minus baseline.
Time Frame: Week 2 and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Number analyzed (Participants) | 176 | 184 | 137
mm Hg
  Baseline | 93.53 (10.24) | 93.81 (11.42) | 94.60 (10.67)
  Change from Baseline | 0.68 (9.58) | -0.58 (10.12) | -1.94 (8.13)
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p = 0.291, ANOVA — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: NEO-OLZ vs NEO-RIS; Test type: Superiority or Other; p = 0.259, ANOVA — [p-value comment as in outcome 8, analysis 1]

16. Secondary Outcome: Vital Signs - Mean Change From Baseline to 10 Week Endpoint in Standing Pulse Rate
Description: Change from Study Period III baseline to endpoint in standing pulse rate. Change = Endpoint minus baseline.
Time Frame: Week 2 and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Number analyzed (Participants) | 175 | 180 | 137
beats per minute
  Baseline | 85.57 (12.83) | 85.32 (13.54) | 82.39 (11.46)
  Change from Baseline | -1.13 (14.20) | -2.05 (13.21) | -0.56 (12.40)
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p = 0.209, ANOVA — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: NEO-OLZ vs NEO-RIS; Test type: Superiority or Other; p = 0.411, ANOVA — [p-value comment as in outcome 8, analysis 1]

17. Secondary Outcome: Vital Signs - Mean Change From Baseline to 10 Week Endpoint in Standing Systolic Blood Pressure
Description: Change from Study Period III baseline to endpoint in standing systolic blood pressure. Change = Endpoint minus baseline.
Time Frame: Week 2 and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Number analyzed (Participants) | 176 | 184 | 137
mm Hg
  Baseline | 123.20 (14.02) | 124.30 (16.23) | 123.20 (13.63)
  Change from Baseline | 0.01 (12.90) | -1.35 (14.22) | -2.36 (10.78)
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p = 0.544, ANOVA — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: NEO-OLZ vs NEO-RIS; Test type: Superiority or Other; p = 0.386, ANOVA — [p-value comment as in outcome 8, analysis 1]

18. Secondary Outcome: Vital Signs - Mean Change From Baseline to 10 Week Endpoint in Body Weight
Description: Change from Study Period III baseline to endpoint in body weight. Change = Endpoint minus baseline.
Time Frame: Week 2 and Week 12
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Number analyzed (Participants) | 179 | 188 | 139
kilograms
  Baseline | 88.28 (23.52) | 90.25 (22.81) | 90.67 (25.39)
  Change from Baseline | 1.85 (3.97) | 1.29 (4.25) | 0.30 (3.26)
Statistical Analysis 1: Comparison: NEO-RIS vs EO-RIS; Test type: Superiority or Other; p = 0.026, ANOVA — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: NEO-OLZ vs NEO-RIS; Test type: Superiority or Other; p = 0.143, ANOVA — [p-value comment as in outcome 8, analysis 1]

ADVERSE EVENTS:
Arm/Group | NEO-OLZ | NEO-RIS | EO-RIS
Serious Adverse Events (participants affected / at risk) | 19/186 | 12/192 | 14/144
Other Adverse Events (participants affected / at risk) | 97 | 100 | 83
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NEO-OLZ (N=186) | NEO-RIS (N=192) | EO-RIS (N=144)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Hallucination, auditory (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
Homicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Hostility (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Paranoia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 3 (3) | 2 (2) | 0 (0)
Schizoaffective disorder (Psychiatric disorders) | 3 (4) | 1 (1) | 0 (0)
Schizophrenia (Psychiatric disorders) | 4 (4) | 1 (1) | 5 (5)
Schizophrenia, paranoid type (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Suicidal ideation (Psychiatric disorders) | 4 (4) | 2 (2) | 4 (4)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | NEO-OLZ | NEO-RIS | EO-RIS
Vision blurred (Eye disorders) | 1/186 (1) | 2/192 (2) | 3/144 (3)
Constipation (Gastrointestinal disorders) | 3/186 (3) | 4/192 (5) | 2/144 (2)
Diarrhoea (Gastrointestinal disorders) | 2/186 (2) | 10/192 (11) | 4/144 (4)
Dry mouth (Gastrointestinal disorders) | 4/186 (4) | 5/192 (6) | 5/144 (5)
Nausea (Gastrointestinal disorders) | 2/186 (2) | 3/192 (3) | 4/144 (4)
Toothache (Gastrointestinal disorders) | 4/186 (4) | 1/192 (1) | 1/144 (1)
Fatigue (General disorders) | 3/186 (3) | 4/192 (4) | 3/144 (3)
Nasopharyngitis (Infections and infestations) | 4/186 (4) | 2/192 (2) | 3/144 (3)
Weight increased (Investigations) | 20/186 (20) | 10/192 (10) | 4/144 (4)
Increased appetite (Metabolism and nutrition disorders) | 5/186 (5) | 9/192 (9) | 3/144 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/186 (1) | 2/192 (2) | 3/144 (3)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1/186 (1) | 2/192 (2) | 6/144 (6)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/186 (0) | 0/192 (0) | 3/144 (3)
Akathisia (Nervous system disorders) | 2/186 (2) | 5/192 (5) | 3/144 (3)
Dizziness (Nervous system disorders) | 3/186 (4) | 4/192 (4) | 1/144 (1)
Extrapyramidal disorder (Nervous system disorders) | 3/186 (3) | 4/192 (4) | 5/144 (5)
Headache (Nervous system disorders) | 9/186 (10) | 8/192 (10) | 7/144 (7)
Hypersomnia (Nervous system disorders) | 1/186 (1) | 0/192 (0) | 3/144 (4)
Lethargy (Nervous system disorders) | 2/186 (2) | 3/192 (3) | 12/144 (13)
Sedation (Nervous system disorders) | 12/186 (13) | 11/192 (11) | 5/144 (5)
Somnolence (Nervous system disorders) | 5/186 (5) | 11/192 (11) | 6/144 (6)
Tremor (Nervous system disorders) | 3/186 (3) | 4/192 (5) | 2/144 (2)
Agitation (Psychiatric disorders) | 3/186 (3) | 3/192 (3) | 3/144 (4)
Anxiety (Psychiatric disorders) | 8/186 (8) | 8/192 (8) | 7/144 (7)
Bruxism (Psychiatric disorders) | 0/186 (0) | 1/192 (1) | 4/144 (4)
Depression (Psychiatric disorders) | 1/186 (1) | 2/192 (2) | 3/144 (3)
Insomnia (Psychiatric disorders) | 7/186 (7) | 16/192 (16) | 4/144 (4)
Restlessness (Psychiatric disorders) | 3/186 (3) | 5/192 (5) | 2/144 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days